CLINICAL TRIAL: NCT03515317
Title: Changes in Cognitive Functions in Patients With Recovery Stage of Traumatic Brain Injury: Effects and Mechanism of Neurofeedback
Brief Title: Effects of Neurofeedback in Cognitive Deficit in Patients With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201704027
Record Dates: First submitted 2018-03-18; First posted 2018-05-03 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Traumatic Brain Injury
Keywords: Cognitive impairments; Low Resolution tomography; Neurofeedback; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LoRETA Z-score NF group (Experimental): BrainMaster Discovery 24E (BrainMaster Technologies, Inc.) combined with Neuroguide software (Applied Neuroscience, Inc.) to conduct both LoRETA Z-score NF. A total treatment dosage of 600 minutes is needed.
  Interventions: Behavioral: LoRETA Z-score NF
- theta/beta NF group (Experimental): BrainMaster Discovery 24E (BrainMaster Technologies, Inc.) combined with Neuroguide software (Applied Neuroscience, Inc.) to conduct both theta/beta NF. A total treatment dosage of 600 minutes is needed.
  Interventions: Behavioral: theta/beta NF
- control group (No Intervention): The control group involves no NF training. The control group will be designed to parallel the cognitive tasks to control for practice effects due to repeated testing (pre- and post- assessments) and the time effect on cognitive function recovery (spontaneous recovery of cognition).

INTERVENTIONS:
Behavioral: LoRETA Z-score NF — LoRETA Z-score NF will be conducted using a 19-lead cap (Electrocap, Inc), which will be placed on the head according to the standard approach of the international 10-20 system with linked ear and ground reference. After the caps will be less than 5 kΩ. During each session, the participants will sit in front of a computer screen on which predesigned games or animations related to the LoRETA Z-score training are played and instructions regarding the inhibitory and reward aspects of the training are taught.
  Arms: LoRETA Z-score NF group
Behavioral: theta/beta NF — The goal of theta/beta NF is to increase the beta power(13-20 Hz) and simultaneously inhibit the theta power (4-8 Hz) relative to a baseline assessed at the beginning of a training session. The electrodes will be placed on Fz and Cz with a linked ear model(A1). The study will use both visual and auditory feedback. Each participant will sit in front of a computer screen on which predesigned games or animations related to the training criteria are played and instructions regarding the inhibitory and reward aspects of the training are taught. The threshold will be set according to 5-min baseline EEG measurements before each session. The thresholds are the mean amplitude of the beta and the theta in 5-min baseline EEG.
  Arms: theta/beta NF group

SUMMARY:
Background: Cognitive impairment is common in patients with traumatic brain injury (TBI) at all levels of severity. Such impairments may affect their ability to return to work and thus increase healthcare costs and the associated economic burdens. Both cognitive rehabilitation and stimulant medications are widely used to manage post-traumatic cognitive impairments; however, previous metaanalyses failed to demonstrate their beneficial effects on cognitive recovery in patients with TBI. Nurses, the first-line healthcare providers, should therefore seek and use an alternative approach for dealing with post-traumatic cognitive deficits.

Purpose: To assess the effects of low resolution tomography (LoRETA) Z -score neurofeedback (NF) and theta/beta NF in alleviating cognitive impairments in patients with TBI as well as the possible mechanism through which they provide this alleviation. We hypothesize that adults with TBI receiving LoRETA Z-score NF and theta/beta NF will experience the improvements in cognitive functions while participants in the control group will not.

DETAILED DESCRIPTION:
Cognitive impairment is the most common and debilitating residual symptom of traumatic brain injury (TBI) at all levels of severity and the prevalence of cognitive impairments varies, depending on the severity of the head injury and the time since the injury. Such impairments substantially affect a person's ability to return to productive activity and health-related quality of life. Furthermore, disabilities related to cognitive impairments following TBI increase healthcare costs and economic burden. Memory, attention, and information processing speed are basic cognitive functions. Deficits in such functions subsequently exacerbate disturbances in more complex cognitive functions (e.g., executive function). Therefore, targeting basic cognitive functions is the first priority of clinical treatments for post-traumatic cognitive impairments.

Cognitive rehabilitation, a nonpharmacological intervention, is the first-line treatment for the management of cognitive impairments following TBI. However, the findings of previous reviews are still debated, with one metaanalysis supporting its beneficial effects on attention recovery and two metaanalyses denying the positive association between cognitive rehabilitation and cognitive recovery. Pharmacotherapies (e.g., methylphenidate) has been potentially used to accelerate cognitive recovery in patients with TBI. Nevertheless, recent systematic reviews failed to prove its effects on cognitive recovery. Moreover, adverse effects may contribute to the discontinuation of stimulant medication use.Taken together, current treatments are insufficient for managing post-traumatic cognitive impairments. Nurses, the first-line healthcare providers, should therefore seek and employ an alternative approach to deal with cognitive impairments following TBI.

Both abnormal network connectivity of the brain (e.g., low neural communication between different brain areas) and dysregulated electroencephalographs (EEGs, e.g., increases in alpha and theta, and decrease in beta) following brain damage have been strongly connected to deficits in memory, sustained attention, and information processing speed. Neurofeedback (NF) can target and alter dysregulated brain functioning by giving real-time feedback of EEG activity to patients. Existing literatures have shown that NF might improve attention performance after TBI. Nonetheless, the effects of NF on other cognitive functions, such as memory and speed of information processing, have not been ascertained. In addition, limited methodological features of previous studies, including single group, pre- and posttreatment study design, small number of participants, and inconsistent treatment protocols, restrict their generalizability and practicability. Most importantly, knowledge regarding cognitive improvements being concomitant with changes in EEGs and the long-term effects of NF on cognitive recovery following TBI is still lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 to 65 years, with a diagnosis of TBI at least 3 months before enrollment(Chronic phase, with an initial Glasgow Coma Scale score of 3-15 (i.e., initially rated in the attention, memory, and information processing speed) by the participants or treating clinician, are able to communicate in Mandarin Chinese, and are able to complete cognitive tasks (having Rancho Los Amigos Scale score>9) will be eligible for inclusion in the study.

Exclusion Criteria:

* The exclusion criteria include premorbid diagnoses of seizures, sleep disorders, psychiatry diseases, substance abuse, and alcoholism. Individuals who are pregnant, in the menopausal transition, and with impairments in vision, hearing, or motor functions that are severe enough to preclude participation in the research will be excluded.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-04-22 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Sustained and selective aspects of visual attention. | three months
  The cognitive functions of the sustained and selective aspects of visual attention assessed by Ruff 2 & 7 Selection Attention Test.
Visual memory function | Three months
  The cognitive functions of visual memory function assessed by Rey Complex Figure Test.
Verbal memory | Three months
  The cognitive functions of verbal memory assessed by Rey Auditory Verbal Learning Test.
Information processing speed. | Three months
  The cognitive functions of information processing speed assessed by Symbol Digit Modalities Test.

SECONDARY OUTCOMES:
Return to productive activity | Three months
  The ability of return to productive measured by the Community integration Questionnaire-Revised (CIQ-R). It is an 18-item ordinal scale designed to assess a person's integration into home and family life, social activity, and productive activity. The home integration, social integration, productivity integration, and electronic social networking subscales have 5, 6, 4, and 3 items, respectively, and each item is scored on a scale of 0 to 2. Higher scores reflect increasing levels of independence.
Health related quality of life | Three months
  The general well-being of individuals and societies, outlining negative and positive features of life, which was evaluated by the quality of life after brain injury (QOLIBRI).The QOLIBRI consists of 37 items covering the following six dimensions of quality of life after TBI: cognition (7 items), self (7 items), daily life and autonomy (7 items), social relationships 6 items), emotions (5 items), and physical problems (5 items). It is scored by a five-point Likert scale with a higher score indicating better quality of life.
Electroencephalography waves | Three month
  Using the BrainMaster Discovery 24E with Neuroguide software.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Taipei Medical University, Taipei
  - Taipei Medical University Hospital., Taipei
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, Taipei
  - Taipei Municipal Wanfang Hospital (managed by Taipei Medical University), Taipei

REFERENCES:
- [Derived] Chen PY, Su IC, Shih CY, Liu YC, Su YK, Wei L, Luh HT, Huang HC, Tsai PS, Fan YC, Chiu HY. Effects of Neurofeedback on Cognitive Function, Productive Activity, and Quality of Life in Patients With Traumatic Brain Injury: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2023 May;37(5):277-287. doi: 10.1177/15459683231170539. Epub 2023 Apr 26. PMID 37125901